CLINICAL TRIAL: NCT05612282
Title: The Impact of the Distribution of Adipose Tissue on the Occurrence of Metabolic Disorders and and the Level of Cardiopulmonary Fitness
Brief Title: The Impact of the Distribution of Adipose Tissue on the Occurrence of Metabolic Disorders and the Level of Cardiopulmonary Fitness
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: N/ST/MN/17/003/3316
Record Dates: First submitted 2022-10-26; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Obesity, Abdominal
Keywords: Adipose tissue; obesity; metabolic disorders
MeSH Terms: conditions — Obesity, Abdominal; Obesity; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- G1a - women: The G1a group consisted of women with obesity, in whom no additional components of the metabolic syndrome were found (n =16)
  Interventions: Diagnostic Test: body composition analysis; Other: anthropometric measurements; Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cardiopulmonary fitness test; Other: nutritional interview
- G1b - men: The G1b group consisted of men with obesity, in whom no additional components of the metabolic syndrome were founds (n =6)
  Interventions: Diagnostic Test: body composition analysis; Other: anthropometric measurements; Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cardiopulmonary fitness test; Other: nutritional interview
- G2a - women: The G2a group consisted of women with obesity, in whom only one additional component of the metabolic syndrome was found (e.g. triglycerides ≥ 150 mg/dl, HDL cholesterol in women < 50 mg/dl, and in men < 40 mg/dl, or glycaemia ≥ 100 mg/dl), but it was not a disease previously diagnosed and treated (n=19)
  Interventions: Diagnostic Test: body composition analysis; Other: anthropometric measurements; Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cardiopulmonary fitness test; Other: nutritional interview
- G2b - men: The G2a group consisted of men with obesity, in whom only one additional component of the metabolic syndrome was found (e.g. triglycerides ≥ 150 mg/dl, HDL cholesterol in women < 50 mg/dl, and in men < 40 mg/dl, or glycaemia ≥ 100 mg/dl), but it was not a disease previously diagnosed and treated (n=11)
  Interventions: Diagnostic Test: body composition analysis; Other: anthropometric measurements; Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cardiopulmonary fitness test; Other: nutritional interview
- G3a - women: Group G3a consisted of women who met the full criteria for diagnosing the metabolic syndrome (n=24)
  Interventions: Diagnostic Test: body composition analysis; Other: anthropometric measurements; Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cardiopulmonary fitness test; Other: nutritional interview
- G3b - men: Group G3a consisted of men who met the full criteria for diagnosing the metabolic syndrome (n=15)
  Interventions: Diagnostic Test: body composition analysis; Other: anthropometric measurements; Other: Interview questionnaire; Diagnostic Test: biochemical parameters; Diagnostic Test: cardiopulmonary fitness test; Other: nutritional interview

INTERVENTIONS:
Diagnostic Test: body composition analysis — A body composition analysis was performed using the bioelectroimpedance method using the Maltron BioScan 920-2 analyzer
Other: anthropometric measurements — An assessment of the status of nutrition based on anthropometric measurements was carried out.
Other: Interview questionnaire — An interview questionnaire concerning the duration of obesity and past diseases was collected. Moreover, the diet and nutritional status were assessed.
Diagnostic Test: biochemical parameters — The concentrations of the following parameters were determined from the blood serum: fasting glucose, fasting insulin, total cholesterol, LDL cholesterol fraction, HDL cholesterol fraction, triglycerides, C-reactive protein (CRP), uric acid, creatinine, and aminotrasferases: alanine (ALT) and aspartate (AST). On the basis of fasting glucose and fasting insulin, the HOMA - IR insulin resistance index was calculated.
Diagnostic Test: cardiopulmonary fitness test — Cardiopulmonary fitness was assessed using the Modified Bruce protocol
Other: nutritional interview — A 7-day nutrition interview was collected. The supply of energy, protein (including amino acids), fat (including fatty acids), carbohydrates, dietary fiber, vitamins and minerals in the usual diet was assessed.

SUMMARY:
The aim of the research was to assess the impact of the distribution of abdominal fat (subcutaneous SAT and visceral VAT estimated at the height of the navel) on selected metabolic parameters and on specific parameters of cardiopulmonary fitness in terms of people with obesity.

DETAILED DESCRIPTION:
The research was carried out in 3 stages. Stage 1 was carried out at the Department of Dietetics and Clinical Nutrition of the UMB. During the visit, the subjects were provided with detailed information concerning the research and every participant signed a voluntary consent to participate in the research. Furthermore, an interview questionnaire concerning the duration of obesity and past diseases was collected, and an assessment of the status of nutrition based on anthropometric measurements was carried out, and a body composition analysis was performed using the bioelectroimpedance method using the Maltron BioScan 920-2 analyzer. Then, patients were issued a referral for laboratory examinations. Stage 2 was carried out at the Medical Laboratory at the University Clinical Hospital in Bialystok, where blood was taken from the ulnar vein (in the amount of 15ml). The concentrations of the following parameters were determined from the blood serum: fasting glucose, fasting insulin, total cholesterol, LDL cholesterol fraction, HDL cholesterol fraction, triglycerides, C-reactive protein (CRP), uric acid, creatinine, and aminotrasferases: alanine (ALT) and aspartate (AST). On the basis of fasting glucose and fasting insulin, the HOMA - IR insulin resistance index was calculated. Stage 3 was carried out at the Maniac Gym Fitness Club in Bialystok, where cardiopulmonary fitness was assessed using the Modified Bruce protocol.

ELIGIBILITY:
Inclusion Criteria:

* primary obesity
* BMI ≥ 30kg/m2 - ≤ 39,99 kg/m2
* gender: women and men
* age: 20-65 lat

Exclusion Criteria:

* secondry obesity
* BMI ≥ 40 kg/m2
* diabetes type 2 or insulin resistance (occurance or treatment)
* endocrine disorders
* eating disorders
* hormonal contraception/hormone replacement therapy
* after steroid therapy
* antiretroviral therapy
* musculoskeletal dysfunctions
* patients after surgery (min 3 months)
* bariatric surgery
* coronary artery disease
* cardiac pacemaker
* pregnancy
* breast - feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research included 91 obese people (59 women and 32 men) who met the criteria for being included in the study and who did not possess exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
The impact of the body compositon parameters (BioScan 920-2) on the risk of metabolic complications of obesity with to use biochemical parameters. | 1 week
  The body weight (kg) was measured using a scale with stadiometer. The height (cm) was measured using a scale with stadiometer. This measurment is needed to calculate BMI (Body Mass Index) and to do a body composition analysis.
  The body composition parameters was determined using the bioimpedance method with a BioScan 920-2 body composition analyzer (Maltron,UK): fat mass (kg), percentage of body fat (%), muscle mass (kg),total body water (kg), basal metabolic rate (kcal).
  Laboratory tests were performed to determine the following serum levels: fasting glucose, fasting insulin, total cholesterol, LDL cholesterol fraction, HDL cholesterol fraction, triglycerides, C-reactive protein (CRP), uric acid, creatinine, and aminotrasferases: alanine (ALT) and aspartate (AST). On the basis of fasting glucose and fasting insulin.
  The HOMA - IR insulin resistance index was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
The impact of the abdominal adipose tissue (VAT, SAT or VAT/SAT) on the risk of metabolic complications of obesity with to use biochemical parameters. | 1 week
  Abdominal adipose tissue was determined using the bioimpedance method with a BioScan 920-2 body composition analyzer (Maltron,UK): visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) and VAT/SAT.
  Laboratory tests were performed to determine the following serum levels: fasting glucose, fasting insulin, total cholesterol, LDL cholesterol fraction, HDL cholesterol fraction, triglycerides, C-reactive protein (CRP), uric acid, creatinine, and aminotrasferases: alanine (ALT) and aspartate (AST). On the basis of fasting glucose and fasting insulin.
  The HOMA - IR insulin resistance index was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
The impact of abdominal adipose tissue distribution (VAT and SAT) on the parameters of cardiopulmonary efficiency. | 1 week
  Abdominal adipose tissue was determined using the bioimpedance method with a BioScan 920-2 body composition analyzer (Maltron,UK): visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) and VAT/SAT.
  Cardiopulmonary fitness was assessed using the Modified Bruce protocol.
Verification of the usefulness of selected anthropometric parameters in the assessment of the risk of developing metabolic disorders in obesity and their relationship with cardiovascular and respiratory efficiency. | 1 week
  An assessment of the status of nutrition based on anthropometric measurements was carried out: body mass index (body weight-kg/weight m2), Waist circumference measurements have been made to the nearest 0.1 centimeter using a tape measure at the uppermost lateral border of the hip crest, Hip circumference was measured at the greater trochanters at the widest part of the hips, Relative fat mass was calculated by the equation: 64-(20 x (height/waist circumference) Laboratory tests were performed to determine the following serum levels: fasting glucose, fasting insulin, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, C-reactive protein (CRP), uric acid, creatinine, and aminotrasferases: alanine and aspartate. On the basis of fasting glucose and fasting insulin The HOMA - IR insulin resistance index was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5 Cardiopulmonary fitness was assessed using the Modified Bruce protocol
The impact of dietary habbits and typicaly diet on on the risk of metabolic complications of obesity with to use biochemical parameters. | 1 week
  An interview questionnaire concerning the duration of obesity and past diseases was collected. Moreover, the diet and nutritional status were assessed.
  A 7-day nutrition interview was collected. The supply of energy, protein (including amino acids), fat (including fatty acids), carbohydrates, dietary fiber, vitamins and minerals in the usual diet was assessed.
  Laboratory tests were performed to determine the following serum levels: fasting glucose, fasting insulin, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, C-reactive protein (CRP), uric acid, creatinine, and aminotrasferases: alanine and aspartate. On the basis of fasting glucose and fasting insulin The HOMA - IR insulin resistance index was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Witczak - Sawczuk, PhD, Study Director — Medical University of Bialystok; Lucyna Ostrowska, Professor, Study Chair — Medical University of Bialystok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mongraw-Chaffin M, Foster MC, Anderson CAM, Burke GL, Haq N, Kalyani RR, Ouyang P, Sibley CT, Tracy R, Woodward M, Vaidya D. Metabolically Healthy Obesity, Transition to Metabolic Syndrome, and Cardiovascular Risk. J Am Coll Cardiol. 2018 May 1;71(17):1857-1865. doi: 10.1016/j.jacc.2018.02.055. PMID 29699611
- [Background] Pimentel Ade C, Scorsatto M, de Oliveira GM, Rosa G, Luiz RR. Characterization of metabolically healthy obese Brazilians and cardiovascular risk prediction. Nutrition. 2015 Jun;31(6):827-33. doi: 10.1016/j.nut.2014.12.024. Epub 2015 Jan 10. PMID 25933489
- [Background] Hoddy KK, Axelrod CL, Mey JT, Hari A, Beyl RA, Blair JB, Dantas WS, Kirwan JP. Insulin resistance persists despite a metabolically healthy obesity phenotype. Obesity (Silver Spring). 2022 Jan;30(1):39-44. doi: 10.1002/oby.23312. Epub 2021 Nov 24. PMID 34816598
- [Background] Perreault M, Zulyniak MA, Badoud F, Stephenson S, Badawi A, Buchholz A, Mutch DM. A distinct fatty acid profile underlies the reduced inflammatory state of metabolically healthy obese individuals. PLoS One. 2014 Feb 10;9(2):e88539. doi: 10.1371/journal.pone.0088539. eCollection 2014. PMID 24520395
- [Background] Kim H, Yoon E, Kim OY, Kim EM. Short-term Effects of Eating Behavior Modification on Metabolic Syndrome-Related Risks in Overweight and Obese Korean Adults. J Obes Metab Syndr. 2022 Mar 30;31(1):70-80. doi: 10.7570/jomes21074. PMID 35296564
- [Background] Zhou YH, Guo Y, Wang F, Zhou CL, Tang CY, Tang HN, Yan DW, Zhou HD. Association of Sex Hormones and Fat Distribution in Men with Different Obese and Metabolic Statuses. Int J Gen Med. 2022 Feb 9;15:1225-1238. doi: 10.2147/IJGM.S351282. eCollection 2022. PMID 35173463
- [Background] Numao S, So R, Matsuo T, Nakagaichi M, Tanaka K. A favorable metabolic profile in metabolically healthy obesity is associated with physical activity level rather than abdominal fat volume in Japanese males. J Phys Ther Sci. 2021 Feb;33(2):137-141. doi: 10.1589/jpts.33.137. Epub 2021 Feb 13. PMID 33642688
- [Background] Matsha TE, Ismail S, Speelman A, Hon GM, Davids S, Erasmus RT, Kengne AP. Visceral and subcutaneous adipose tissue association with metabolic syndrome and its components in a South African population. Clin Nutr ESPEN. 2019 Aug;32:76-81. doi: 10.1016/j.clnesp.2019.04.010. Epub 2019 Jun 3. PMID 31221294
- [Background] Osorio-Conles O, Vega-Beyhart A, Ibarzabal A, Balibrea JM, Vidal J, de Hollanda A. Biological Determinants of Metabolic Syndrome in Visceral and Subcutaneous Adipose Tissue from Severely Obese Women. Int J Mol Sci. 2022 Feb 21;23(4):2394. doi: 10.3390/ijms23042394. PMID 35216509
- [Background] Schorr M, Dichtel LE, Gerweck AV, Valera RD, Torriani M, Miller KK, Bredella MA. Sex differences in body composition and association with cardiometabolic risk. Biol Sex Differ. 2018 Jun 27;9(1):28. doi: 10.1186/s13293-018-0189-3. PMID 29950175
- [Background] Chashmniam S, Hashemi Madani N, Nobakht Mothlagh Ghoochani BF, Safari-Alighiarloo N, Khamseh ME. The metabolome profiling of obese and non-obese individuals: Metabolically healthy obese and unhealthy non-obese paradox. Iran J Basic Med Sci. 2020 Feb;23(2):186-194. doi: 10.22038/IJBMS.2019.37885.9004. PMID 32405361
- [Background] Kaess BM, Pedley A, Massaro JM, Murabito J, Hoffmann U, Fox CS. The ratio of visceral to subcutaneous fat, a metric of body fat distribution, is a unique correlate of cardiometabolic risk. Diabetologia. 2012 Oct;55(10):2622-2630. doi: 10.1007/s00125-012-2639-5. Epub 2012 Aug 17. PMID 22898763